CLINICAL TRIAL: NCT03698071
Title: Soluble CD95 Ligand Role in the Pathophysiology of ANCA Associated Vasculitis
Brief Title: Soluble CD95 Ligand Role in the Pathophysiology of Antineutrophil Cytoplasmic Antibody (ANCA) Associated Vasculitis
Acronym: VASC-FAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2018/22
Record Dates: First submitted 2018-10-04; First posted 2018-10-05 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: ANCA Associated Vasculitis
Keywords: ANCA associated vasculitis; Granulomatosis with polyangiitis; microscopic polyangiitis; eosinophilic granulomatosis with polyangiitis; soluble-CD95-Ligand
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Churg-Strauss Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ANCA associated vasculitis (Experimental)
  Interventions: Biological: blood sample; Biological: urine sample

INTERVENTIONS:
Biological: blood sample — 30 ml whole blood for Peripheral blood mononuclear cell (PBMC) and monocytes isolation
Biological: urine sample — 6 ml

SUMMARY:
The study aims at defining the role of soluble CD95 Ligand in the physiopathology of a rare group of inflammatory diseases: ANCA associated vasculitis. Soluble CD95 Ligand might have a prognostic and diagnostic interest as well as potential for the discovery of new therapeutic strategies.

DETAILED DESCRIPTION:
ANCA associated vasculitis are a rare group of diseases and potentially life-threatening inflammatory conditions. There is an urgent need to describe prognostic factors and to discover new therapeutic pathways. Soluble CD95-L is a cleaved part of CD95-L which binds the CD95 Death receptor. s-CD95-L has pro-inflammatory properties for Th17 lymphocytes and Neutrophils, two cells implicated in ANCA associated vasculitis. It also plays a role in systemic lupus erythematosus (which present with the same type of renal glomerulonephritis as ANCA-associated vasculitis). Finally, it has already be found elevated in this group of diseases. The investigators hypothesized that s-CD95-L levels might be a prognostic factor in ANCA associated vasculitis and the study of the molecular mechanisms involved could provide new therapeutic targets.

The study will recruit 50 patients with ANCA associated vasculitis followed in Bordeaux University Hospital. Among classical disease activity information, blood and urine samples will be collected at each visit to study s-CD95-L. Fundamental research will be realized on patients' sample to study molecular mechanisms involved.

Clinical and biological disease activity, treatment and outcomes will be studied in correlation with s-CD95-L to describe their potential prognostic role. Patients will be followed at regular intervals, as their usual follow-up would request. No extra visit will be needed and blood samples will be drawn at the same time as those drawn for clinical purposes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ANCA associated vasculitis according to the Chapel-Hill Consensus Conference - 2012 modified version
* Age ≥ 18 years
* being affiliated to health insurance
* willing to participate and to sign informed consent.

Exclusion Criteria:

* Pregnant or breastfeeding women,
* patient concerned by articles L 1121-5 to L 1121-8 (persons deprived of their liberty by a judicial or administrative decision, minors, persons of legal age who are the object of a legal protection measure or unable to express their consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-09-18 (Actual)

PRIMARY OUTCOMES:
Change of quantitative levels of s-CD95-L in ANCA associated vasculitis between baseline and Month 12 | At baseline (Day 0) and 12 months from baseline

SECONDARY OUTCOMES:
Change of disease activity scores for ANCA associated vasculitis between baseline and Month 12 | At baseline (Day 0) and 12 months from baseline
  Birmingham Vasculitis Activity Score - Version 3 (BVAS 3.0) The Birmingham Vasculitis Activity Score (BVAS) is a method for assessing the activity of vasculitis. Note that scoring ranges are higher when any of the features are new or worse. Creatinine levels can be scored at patient's first assessment only. The maximum score is 63 points for present symptoms and 32 points for new symptoms or symptoms which had worsened within the previous weeks.
Change of disease activity scores for ANCA associated vasculitis between baseline and Month 12 | At baseline (Day 0) and 12 months from baseline
  Vasculitis Damage Index (VDI)
Change of quantification of s-CD95-L in the blood and urine samples of ANCA associated vasculitis between baseline and Month 12 | At baseline (Day 0) and 12 months from baseline
Change of quantification of ANCA in the blood samples of ANCA associated vasculitis between baseline and Month 12 | At baseline (Day 0) and 12 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Patrick BLANCO, Prof, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux - Service d'Immunologie et Immunogénétique, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No